CLINICAL TRIAL: NCT01928914
Title: A Randomized, Placebo-Controlled Study to Evaluate the Effect of Tafenoquine (SB252263) on the Electrocardiogram (ECG) With Focus on Cardiac Repolarization (QTc Duration) in Healthy Subjects
Brief Title: Tafenoquine Thorough QTc Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 114582
Record Dates: First submitted 2012-03-29; First posted 2013-08-27 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Malaria, Vivax
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Placebo Comparator): Subjects in group 1 receive placebo for tafenoquine and placebo for moxifloxacin on three consecutive days of dosing
  Interventions: Drug: Placebo for Tafenoquine; Drug: Placebo for moxifloxaxin
- Group 2 (Experimental): Subjects in group 2 receive 400mg of tafenoquine and placebo for moxifloxacin on three consecutive days of dosing
  Interventions: Drug: Tafenoquine 1200mg; Drug: Placebo for Tafenoquine
- Group 3 (Active Comparator): Subjects in group 1 receive placebo for tafenoquine and placebo for moxifloxacin on days 1 and 2. On day 3, subjects receive placebo for tafenoquine and 400mg moxifloxacin.
  Interventions: Drug: moxifloxacin; Drug: Placebo for Tafenoquine; Drug: Placebo for moxifloxaxin
- Group 4 (Experimental): Subjects in group 1 receive placebo for tafenoquine and placebo for moxifloxacin on days 1 and 2. On day 3, subjects receive placebo for moxifloxacin and 300mg of tafenoquine
  Interventions: Drug: Tafenoquine 300mg; Drug: Placebo for Tafenoquine; Drug: Placebo for moxifloxaxin
- Group 5 (Experimental): Subjects in group 1 receive placebo for tafenoquine and placebo for moxifloxacin on days 1 and 2. On day 3, subjects receive placebo for moxifloxacin and 600mg of tafenoquine
  Interventions: Drug: Tafenoquine 600mg; Drug: Placebo for Tafenoquine; Drug: Placebo for moxifloxaxin

INTERVENTIONS:
Drug: Tafenoquine 300mg — Single dose of Tafenoquine give on Day 3 only
  Arms: Group 4
Drug: Tafenoquine 600mg — Single dose of Tafenoquine given on Day 3 only
  Arms: Group 5
Drug: Tafenoquine 1200mg — 400mg Dose of Tafenoquine given on each of the three consecutive dosing days
  Arms: Group 2
Drug: moxifloxacin — moxifloxacine given on Day 3 only
  Arms: Group 3
Drug: Placebo for Tafenoquine — Placebo given on all three days to all groups except for group 5 on Day 3
Drug: Placebo for moxifloxaxin — Placebo for moxifloxacin, given to all groups on all days except for Group 3 on Day 3
  Arms: Group 1; Group 3; Group 4; Group 5

SUMMARY:
This will be a randomized, single-blind, placebo controlled, parallel group study. Approximately 260 subjects will be enrolled in five groups. This study is designed to compare the effects of tafenoquine, administered as single dose as well as administered over three consecutive days, on the changes in QT duration to those observed in subjects dosed with either moxifloxacin or placebo.

DETAILED DESCRIPTION:
SB-252263 (tafenoquine, TQ) is a new 8-aminoquinoline antimalarial drug being developed by GlaxoSmithKline (GSK) and the Medicines for Malaria Venture with the assistance and historical support of the Walter Reed Army Institute of Research. Tafenoquine has been shown to be effective in the treatment of plasmodial infections in vitro, in pre-clinical models in vivo, and during early phase clinical studies for radical cure and eradication of liver hypnozoites in patients infected with Plasmodium vivax. This study is designed to compare the effects of tafenoquine mono-therapy, administered as a single dose or administered on 3 consecutive days, on the changes in QT duration to those observed in subjects dosed with either Avelox (moxifloxacin hydrochloride) or placebo. This will be a randomized, single-blind, placebo controlled, parallel group study. Parallel group design is chosen because tafenoquine has a long half-life, about 14 to 19 days, and therefore a cross-over design is not a practical alternative. Moxifloxacin will be used as a positive control in order to validate the sensitivity of the study in detecting QTc change. Moxifloxacin has been shown to prolong the QT interval in a dose-dependent manner in patients and healthy volunteers, and the QTc prolongation has been well quantified.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and baseline ECG cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 90 days post-last dose.
* Body weight ≥50 kg for men and ≥45 kg for women and BMI within the range 18.5 to 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Documented Glucose-6-phosphate dehydrogenase (G6PD) deficiency, determined by a quantitative assay of enzyme activity.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of thalassaemia; or current or past history of methemoglobinemia or methemoglobin percentage above the reference range at screening.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of 2nd degree or higher AV block.
* Donation of blood or blood products in excess of 500 mL within a 56 day period prior to enrolment.
* Subjects with a hemoglobin values outside the normal range. A single repeat is allowed for eligibility determination.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination)
* PR Interval <120 and >220 msec
* QRS Duration <70 and >120 msec
* QTc, QTcB or QTcF Interval >450 msec
* Heart Rate, for male subjects <45 and >100 bpm, and for female subjects <50 and >100 bpm
* Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolff Parkinson White [WPW] syndrome).
* Sinus Pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (>3 consecutive ventricular ectopic beats).
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80o proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Pregnant females as determined by positive (serum or urine) hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-07-26 (Actual); Primary Completion 2012-06-04 (Actual); Study Completion 2012-06-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF for 1200 mg dose of tafenoquine compared to baseline | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  Contineous QTcF will be electronically recorded using holtor monitors. The primary comparison of interest is the mean time-matched change from baseline in QTcF for the difference tafenoquine-placebo for 1200mg dose of tafenoquine at each timepoint.

SECONDARY OUTCOMES:
Change from Baseline in QTcB, QTcI, QT, and HR for 1200mg dose of tafenoquine | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  electronic ECGs collected using holter monitors will be analysed to measure QTcF QTcB, QTcI, QT, and Heart Rate (HR)
Change from Baseline in QTcF QTcB, QTcI, QT, and HR for 300 mg single dose of tafenoquine | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  electronic ECGs collected using holter monitors will be analysed to measure QTcF QTcB, QTcI, QT, and Heart Rate (HR)
Change from Baseline in QTcF, QTcB, QTcI, QT, and HR for placebo | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  electronic ECGs collected using holter monitors will be analysed to measure QTcF QTcB, QTcI, QT, and Heart Rate (HR)
Change from Baseline in QTcF, QTcB, QTcI, QT, and HR for moxifloxacin | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  electronic ECGs collected using holter monitors will be analysed to measure QTcF QTcB, QTcI, QT, and Heart Rate (HR)
Plasma concentrations and derived pharmacokinetic parameters AUC(0-t), Cmax, and tmax of tafenoquine | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  Blood samples will be collected at pre-dose on Days 1 and 2, and Day 3: pre-dose, 1, 2, 3, 4, 5, 6, 9, 12, 15, 20, 24, 36, 48 and 72 hours post Day 3 dose, to measure plasma concentrations and derived pharmacokinetic parameters AUC(0-t), Cmax, and tmax of tafenoquine
Safety and tolerability of tafenoquine as assessed by 12-lead ECGs, vital signs, adverse events, and clinical laboratory tests | Day 1, Day 2 and Day 3
  Safety and tolerability of tafenoquine as assessed by 12-lead ECGs, vital signs, adverse events, and clinical laboratory tests
Change from Baseline in QTcF QTcB, QTcI, QT, and HR for 600 mg single dose of tafenoquine | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  electronic ECGs collected using holter monitors will be analysed to measure QTcF QTcB, QTcI, QT, and Heart Rate (HR)
Plasma concentrations and derived pharmacokinetic parameters AUC(0-t), Cmax, and tmax of moxifloxacin | Day 1, Day 2, day 3, Day 4, Day 5 and Day 6
  Blood samples will be collected at pre-dose on Days 1 and 2, and Day 3: pre-dose, 1, 2, 3, 4, 5, 6, 9, 12, 15, 20, 24, 36, 48 and 72 hours post Day 3 dose, to measure plasma concentrations and derived pharmacokinetic parameters AUC(0-t), Cmax, and tmax of moxifloxacin

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Culver City, California
  - GSK Investigational Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 114582 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114582?search=study&study_ids=114582#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114582 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register